CLINICAL TRIAL: NCT06660940
Title: A Randomized, Double-blind, Multicenter Clinical Trial of Keluoxin Capsules in the Treatment of Diabetic Kidney Disease with Diabetic Retinopathy
Brief Title: Clinical Trial of Keluoxin Capsules in the Treatment of Diabetic Kidney Disease with Diabetic Retinopathy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BOJI2022080XY
Record Dates: First submitted 2024-10-21; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Kidney Disease; Diabetic Retinopathy
Keywords: Diabetic kidney disease; Keluoxin Capsules; Diabetic retinopathy
MeSH Terms: conditions — Diabetic Nephropathies; Diabetic Retinopathy | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Keluoxin Capsules (Experimental): Patients will take Keluoxin Capsules and renin-angiotensin-aldosterone system inhibitors (RAASIs).
  Interventions: Drug: Keluoxin Capsules; Drug: Irbesartan
- Placebo (Placebo Comparator): Patients will take placebo and RAASIs.
  Interventions: Drug: Keluoxin Capsule Simulants; Drug: Irbesartan

INTERVENTIONS:
Drug: Keluoxin Capsules — Treatment period (52 weeks):Keluoxin Capsules, 4 capsules/time, swallow with warm water after meals, 3 times/day
  Arms: Keluoxin Capsules
Drug: Keluoxin Capsule Simulants — Treatment period (52 weeks):Keluoxin Capsule Simulants, 4 capsules/time, swallow with warm water after meals, 3 times/day
  Arms: Placebo
Drug: Irbesartan — 1. Lead-in period (2-4 weeks): Irbesartan 75-300mg/d, QD;
  2. Treatment period (52 weeks): Irbesartan 75-300mg/d, QD

SUMMARY:
The purpose of the study is to evaluate the efficacy of Keluoxin Capsules for the treatment of diabetic kidney disease (DKD) and diabetic retinopathy (DR) compared to placebo on a conventional treatment basis.

DETAILED DESCRIPTION:
DKD and DR are the main microvascular complications of diabetes mellitus. DKD is currently the leading cause of end-stage renal disease (ESRD), while DR is the leading cause of blindness in the working age population. DKD and DR have similar pathogenesis and pathological manifestations. For patients with DKD whose estimated glomerular filtration rate (eGFR) ≥ 30ml/min/1.73m2, the proportion of patients with mild, moderate and severe non-proliferative diabetic retinopathy (NPDR) and proliferative diabetic retinopathy (PDR) was 17.38%, 27.57%, 12.29% and 2.28%, respectively. The previous research results showed that Keluoxin Capsules could improve DKD symptoms, reduce proteinuria, protect renal function, and stabilize or improve DR. This study is a multicenter,double-blind, randomized controlled trial. We plan to enroll 460 participants, who will be randomized to receive either Keluoxin capsules(230 cases) or placebo(230 cases) on a conventional treatment basis for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old, either sex;
* Meeting the diagnostic criteria for type 2 diabetes mellitus and DKD;
* The target eye met the diagnostic criteria for type 2 DR and the fundus showed moderate or severe NPDR;
* Have been treated with an adequate dose of RAASIs for more than 4 weeks;
* The 24h UTP between 0.5g and 3.5g (results of two tests);
* The eGFR ≥30ml/min/1.73m2；
* Blood pressure (BP) ≤ 140/90mmHg;
* Hemoglobin A1c (HbA1c) < 9%;
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients with a known or suspected history of allergy to the test drug and its excipients;
* Various primary kidney diseases or non-diabetic kidney disease as judged by the investigator;
* Heat-toxin syndrome: swelling and pain the throat , redness, swelling, and pain in the eyes, mouth and tongue sores, swollen and painful gums, cough with yellow phlegm, stool stem nod, deep colored urine, red tongue with yellow coating; cold-dampness syndrome: poor appetite, borborygmus, diarrhoea, drowsiness, clear urine in large amounts and high frequency, menstrual disorders, aversion to cold and cold limbs; meet the either manifestation of heat-toxin syndrome or cold-dampness syndrome, that is, the need to be excluded;
* The patient's eye has any of the following conditions:

  1.Target eye (if both eyes of the patient meet the inclusion criteria, the target eye will be determined by the investigator from a medical point of view. In principle, the eye with more severe lesion will be chosen as the target eye, and the eye with clearer refractive media will be chosen if the lesions are of the same degree):
  1. Received periocular corticosteroid injections within 3 months prior to screening;
  2. Use of Chinese patent medicines or chemical drugs with therapeutic effects on DR (e.g., Calcium Dobesilate, Difrarel, Qiming Granules, Shuangdan Mingmu Capsules) within 2 weeks prior to screening;
  3. Suffering from other retinal diseases affecting the macula, e.g. central retinal vein occlusion (CRVO), branch retinal vein occlusion (BRVO), wet age-related macular degeneration (AMD), choroidal neovascularization (CNV), CI-DME, ocular ischemic syndrome, Irvine-Gass syndrome, radiation retinopathy;
  4. Suffering from other eye diseases that affect vision, such as glaucoma, uveitis, optic neuropathy, retinal detachment;
  5. Have undergone the following ophthalmic surgeries or treatments: vitrectomy, macular buckling, glaucoma filtration surgery, panretinal photocoagulation, macular photocoagulation, photodynamic therapy, optic neurotomy, optic nerve sheath fenestration, etc;
  6. Undergone the following eye surgeries within 3 months prior to screening, including cataract surgery and keratoplasty;
  7. The need for cataract surgery during the study period;
  8. Presence of refractive medium opacity and/or pupillary abnormality that affect fundus photography and OCTA imaging; 2. Either eye:

  <!-- -->

  1. Received intravitreal injection of anti-vascular endothelial growth factor (VEGF) drugs or corticosteroids within 3 months prior to screening;
  2. Suffering from active inflammation of the eye or periocular area (e.g., hordeolum, infectious conjunctivitis, keratitis, scleritis, endophthalmitis);
  3. Suffering from intraocular or intraorbital space-occupying lesions, and malignancy cannot be excluded.
* Have a history of using systemic glucocorticoids and immunosuppressants within 3 months prior to enrolment;
* Experienced active bleeding within 3 months prior to enrolment;
* The eGFR decreased by ≥ 30% within 3 months prior to enrolment;
* Patients with a history of unilateral or bilateral renal artery stenosis;
* BP < 90/60 mmHg;
* Serious acute complications of diabetes mellitus, serious infections within 4 weeks prior to enrolment;
* Serum albumin (ALB) < 30g/L, hemoglobin ≤ 90g/L;
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) reaches more than two times of the upper limit of normal level;
* Comorbid with serious diseases of other organs such as cardiovascular disease, respiratory disease, and other serious diseases that may affect the patient's life;
* Patients with malignancy or malignant diseases that affect the overall prognosis;
* Pregnant and lactating women or women with childbearing plans within 6 months;
* Those who have participated in a clinical trial of another drug within 3 months prior to randomization (referring to those who are randomized and treated with the trial drug);
* Others who were judged by the investigator to be inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The 24-hour urinary protein quantitation (24h UTP) level and changes from baseline at 52 weeks. | baseline,52 weeks
  Differences between groups using the changes in 24h UTP relative to baseline after 52 weeks treatment.
The macular vascular density or foveal avascular zone area and changes from baseline at 52 weeks. | baseline,52 weeks
  Differences between groups using the changes in macular vascular density or foveal avascular zone area relative to baseline after 52weeks treatment.

SECONDARY OUTCOMES:
The urine albumin creatine ratio (UACR) level and changes from baseline at each visit. | baseline, 8, 16, 28, 40, and 52 weeks
  Differences between groups using the changes in UACR relative to baseline after 8, 16, 28, 40, and 52 weeks treatment.
The eGFR level and changes from baseline at each visit. | baseline, 8, 16, 28, 40, and 52 weeks
  Differences between groups using the changes in eGFR relative to baseline after 8, 16, 28, 40, and 52 weeks treatment.
The ophthalmic indicators level and changes from baseline at each visit. | baseline, 8, 16, 28, 40, and 52 weeks
  Differences between groups using the changes in ophthalmic indicators (macular perfusion density, foveal avascular zone acircularity index, macular thickness, et al) relative to baseline after 8, 16, 28, 40, and 52 weeks treatment.
The Chinese medicine syndrome scores and changes from baseline at each visit. | baseline, 8, 16, 28, 40, and 52 weeks
  Differences between groups using the changes in Chinese medicine syndrome scores relative to baseline after 8, 16, 28, 40, and 52 weeks treatment. (The score of the Chinese medicine syndrome scale ranges from 0 to 24, with higher scores mean a worse outcome.)
The diabetes quality of life measure (DQOL) scale (each domain score) and changes from baseline at each visit. | baseline, 8, 16, 28, 40, and 52 weeks
  Differences between groups using the changes in DQOL scale (each dmain score) relative to baseline after 8, 16, 28, 40, and 52 weeks treatment.
Proportions of patients with serum creatinine doubling | baseline, 8, 16, 28, 40, and 52 weeks
  Differences between groups using the proportions of patients with serum creatinine doubling at each visit.
Proportions of patients with progressed to ESRD | baseline, 8, 16, 28, 40, and 52 weeks
  Differences between groups using the proportions of patients with progressed to ESRD at each visit.
eGFR decline slope | baseline, 8, 16, 28, 40, and 52 weeks
  Differences between groups using the eGFR decline slope after 8, 16, 28, 40, and 52 weeks treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei chen, Principal Investigator — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No